CLINICAL TRIAL: NCT04441229
Title: A Prospective, Observational Study of Mobile Attentional Bias Modification Training (ABMT) in the Pediatric Multiple Sclerosis (MS) Population
Brief Title: Mobile Attentional Bias Modification Training in Pediatric MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00810
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Pediatric Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Patients age 12-24 diagnosed with pediatric-onset Multiple Sclerosis
  Interventions: Behavioral: ABMT mobile application

INTERVENTIONS:
Behavioral: ABMT mobile application — After consent/assent, participants will complete 1 hour-long, in-person or remote, baseline study visit at the Multiple Sclerosis Comprehensive Care Center. During this visit, participants will complete baseline study surveys and a brief computerized attention bias assessment and be trained on the use of the ABMT mobile application. Participants will then complete at-home game play 4 days a week, for 30 days, using an iOS mobile device, approximately 10-15 minutes each day. Subjects will complete weekly online study surveys via REDCap or MyCap (Mobile REDCap Application). At the conclusion of participation, participants will complete online end of study surveys via REDCap or MyCap.
  Parents of participants will complete surveys at the baseline visit, followed by online surveys at Week 2 and at the end of study. For participants who are 18 years old or older, parental participation will not be required.

SUMMARY:
This study will examine the feasibility of using a mobile ABMT application as a treatment modality in the Pediatric Multiple Sclerosis population. Participants will be asked to undergo one hour-long baseline evaluation, followed by at-home ABMT application sessions. Subjects will complete online REDCap or MyCap surveys weekly and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-24 years
* Confirmed Diagnosis of Multiple Sclerosis with onset < 17 years and 11 months (defined by the 2013 International Pediatric MS Study Group (IPMSSG) criteria (Krupp, Tardieu, Amato, Banwell, Chitnis, Dale, Ghezzi, Hintzen, Kornberg, Pohl, Rostasy, Tenembaum, Wassmer, & Sclerosis, 2013) and the 2010 McDonald criteria (Polman et al., 2011).)
* Followed at NYU Multiple Sclerosis Comprehensive Care Center
* Access to a mobile device with iOS (devices will be provided to subjects if this criteria is not met, see section 4.4)
* Active or concurrently enrolled in the ongoing US Network of Pediatric MS Centers Study Consortium

Exclusion Criteria:

* Previous report of an IQ < 70
* Wide-Range Achievement Test-Fourth Edition (Wilkerson, 2006) Reading Subtest standard score <85
* Non-English speaking, learned English in the past three years, or learned English after the age of 12 years
* Not willing to comply with all study procedures
* Insufficient visual and motor ability to operate the intervention and assessments

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Proportion of "compliant" participants | 30 days
  Individuals will be categorized as "compliant" if they interact with the mobile ABMT a minimum of 3 times per week for a minimum of three of the four weeks across the study period of 30 days. We will consider reaching 50% of compliant participants to indicate that the intervention is feasible for continued study. Descriptive analyses will be completed to identify any trends in predicting those participants who are most likely to be compliant (ie. age, gender, baseline function).

SECONDARY OUTCOMES:
Preliminary efficacy composite score | 3 months
  Investigators convert performance at baseline and study end across study measures SCARED P/C,CDI-II, MASC-2, BDI-II, BAI, and PANAS to scaled age normative scores. Differences in scaled scores, indicating change following intervention, will be calculated for each compliant participant (defined as above) and averaged for group metrics. Descriptive analyses will be completed to identify any trends in predicting those participants who are most likely to have improvement in anxiety and mood at study end (ie., age, gender, baseline function) as well as corresponding degree of use of the mobile ABMT with magnitude of benefit.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: leigh.charvet@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to leigh.charvet@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.